CLINICAL TRIAL: NCT04693442
Title: A Multi-centre, Prospective Study to Examine the Relationship Between Neutrophil Function and Sepsis in Adults and Children With Severe Thermal Injuries
Brief Title: Relationship Between Neutrophil Function and Sepsis in Adults and Children With Severe Thermal Injuries
Acronym: SIFTI-2
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital Birmingham NHS Foundation Trust (Other)
Collaborators: The Scar Free Foundation (Unknown); University of Birmingham (Other)
Responsible Party: Principal Investigator, Naiem Moiemen, Burns and Plastics Consultant, University Hospital Birmingham NHS Foundation Trust
Other Study IDs: RRK5814; IRAS Project ID 200366 (Other: HRA)
Record Dates: First submitted 2019-04-16; First posted 2021-01-05 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2020-12

CONDITIONS: Burns
MeSH Terms: conditions — Burns | interventions — Urination; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — skin tissue, serum, plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Burn patients: with the condition
  Interventions: Other: taking of blood, urine and blood samples and objective scar assessment
- Control group: without the condition (blood sampling only for adults) and children undergoing general anaesthetic procedures that involve skin resections (blood sampling and excised skin)

INTERVENTIONS:
Other: taking of blood, urine and blood samples and objective scar assessment — blood, urine and skin tissue sampling & scar assessment questionnaires
  Groups: Burn patients

SUMMARY:
The study aims to validate neutrophil function, immature granulocyte and plasma free DNA levels as predictive diagnostic biomarkers of sepsis in burn patients. Inclusion criteria includes healthy volunteers, patients aged 5-15 years old with burns affecting 20% or less Total Body Surface Area (TBSA) and patients aged 16 or above with burns affecting >15% TBSA. The study involves taking blood, tissue and urine samples.

DETAILED DESCRIPTION:
The initial cohort for SIFTI-2 will be generated from patients attending the Birmingham Burns Centre at Queen Elizabeth Hospital Birmingham (QEHB) and Birmingham Children's Hospital (BCH). The cohort will be comprised of patients with moderate and severe burns (injury to more than 15% of the body surface area [TBSA] in adults and 20% TBSA in children). The investigators currently treat between 30-40 patients in this category each year. In order to thoroughly characterise the longitudinal neutrophil response to burn injury and to investigate its potential relationship with outcome post-burn, the ivestigators will measure the genomic, phenotypic and functional response of peripheral blood neutrophils across time in burn-injured patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 1-15 years admitted with a ≥20%TBSA
* Patients aged 16 and over admitted with a ≥15% TBSA
* Patients presented within 24 hours of thermal injury

Exclusion Criteria:

* Associated multiple injuries with Injury severity score > 25
* Decision not to treat made on admission due to the severity of the injury
* Patients with chemical and deep electrical burns
* Premorbid conditions
* Active Malignancy
* Patients receiving glucocorticoid treatment
* Multiple limb amputations
* Patients with known long term infections (i.e., Hepatitis B & C, Human Immune Deficiency [HIV])

Ages: 1 Year to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Subjects will be admitted to any Burn Centre participating in the study. This includes but not limited to:
  Queen Elizabeth Hospital Birmingham; Birmingham Children's Hospital; Mid Essex NHS Trust, Broomfield Hospital, Chelmsford
  The patients will be new burns patients presented within 24 hours of thermal injury. They will be identified by the admitting doctor from the Burns Team.
Sampling Method: Probability Sample
Enrollment: 245 (Estimated)
Dates: Start 2016-11-18 (Actual); Primary Completion 2022-01-31 (Estimated); Study Completion 2022-01-31 (Estimated)

PRIMARY OUTCOMES:
Diagnosis of sepsis | 2 years
  Sepsis will be evaluated according to the 2007 American Burn Association (ABA) diagnostic criteria for sepsis in burns. Specifically, sepsis will be diagnosed when 3 of the following criteria are met along with a positive bacterial culture or when evidence of a clinical response to antibiotics is detected:
  1. Temperature (>39°C or <36°C)
  2. progressive tachycardia (>110 beats per minute
  3. progressive tachypnea (>25 breaths per minute not ventilated or minute ventilation >12 L/minute ventilated)
  4. thrombocytopenia (<100,000/μl; not applied until 3 days after initial resuscitation)
  5. hyperglycaemia (untreated plasma glucose >200 mg/dl, >7 units of insulin/hr intravenous drip, or >25% increase in insulin requirements over 24 hours)
  6. feed intolerance >24 hours (abdominal distension, residuals two times the feeding rate, or diarrhoea >2500 ml/day)

SECONDARY OUTCOMES:
In-hospital mortality | 2 years
  Death while in-hospital
Predictive mortality scores | 2 years
  Predictive mortality scores are measured by Revised Baux Score, Abbreviated Burn Severity Index (ABSI), and APACHE II
Multiple Organ Failure/dysfunction syndrome (MOF/MODS) | 2 years
  The presence of altered organ function where homeostasis cannot be maintained without intervention using Denver 2 and SOFA scores. For Denver score, MOF is defined as > 3, two (2) organ system involved for 2 consecutive days while in SOFA, MOF> = 4 , two (2) organ system involved for first 24 hours. In the subsequent time points, only cardiac scores for SOFA and Denver 2 are recorded.
Thromboembolic complications | 2 years
  Clinical signs and symptoms associated with thrombosis, i.e., pulmonary embolism, deep vein thrombosis. Clinical investigation to confirm thrombosis will be based on any of the following imaging procedure: CTPA, VQ Scan, USS, Venogram, D-dimer results
Vancouver Scar Scale (VSS) | 2 years
  This scale uses a numerical assessment of four skin characteristics including: Height (range, 0-4), Pliability (range, 0-4), Vascularity (range, 0-3), and Pigmentation (range, 0-3). The assessors choose a numerical value for each of these characteristics based on a comparison with normal skin.
Patient and Observer Scar Assessment Scale | 2 years
  Patient and Observer Scar Assessment Scale (POSAS, version 2.0) - The POSAS questionnaire seeks to measure scar quality and is a subjective scar scale that consists of two parts: a Patient Scale and an Observer Scale. Both scales contain six items that are scored numerically on a ten-step scale and together they make up the 'Total Score' of the Patient and Observer Scale. The POSAS Patient scale assesses the scar in terms of pain, itching, scar colour, stiffness, thickness and irregularity and overall opinion. The POSAS Observer scale assesses the scar in terms of vascularity, pigmentation, thickness, relief, pliability, surface area and overall opinion.
Brisbane Burn Scar Impact Profile | 2 years
  Brisbane Burn Scar Impact Profile (BBSIP, version 1.0) - This questionnaire assesses the health-related quality of life in people with burn scars. It consists of seven parts which measure; (a) the overall impact of burn scars (itch, pain and other sensations, and their impact on the subject), (b) the impact of the burn scars on work and daily activities, (c) the impact of the burn scars on relationships and social interactions, (d) the subjects perception of the impact of the burn scars on their appearance, (e) the subjects emotional reactions towards their scars and (f) the physical symptoms caused by the burn scars.

CONTACTS AND LOCATIONS:
Overall Officials: Naiem Moiemen, Surgeon, Principal Investigator — The Scar Free Foundation
Locations (1):
- University Hospitals Birmingham NHS Foundation Trust, Birmingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Farina JA Jr, Rosique MJ, Rosique RG. Curbing inflammation in burn patients. Int J Inflam. 2013;2013:715645. doi: 10.1155/2013/715645. Epub 2013 May 20. PMID 23762773
- [Background] Xiao W, Mindrinos MN, Seok J, Cuschieri J, Cuenca AG, Gao H, Hayden DL, Hennessy L, Moore EE, Minei JP, Bankey PE, Johnson JL, Sperry J, Nathens AB, Billiar TR, West MA, Brownstein BH, Mason PH, Baker HV, Finnerty CC, Jeschke MG, Lopez MC, Klein MB, Gamelli RL, Gibran NS, Arnoldo B, Xu W, Zhang Y, Calvano SE, McDonald-Smith GP, Schoenfeld DA, Storey JD, Cobb JP, Warren HS, Moldawer LL, Herndon DN, Lowry SF, Maier RV, Davis RW, Tompkins RG; Inflammation and Host Response to Injury Large-Scale Collaborative Research Program. A genomic storm in critically injured humans. J Exp Med. 2011 Dec 19;208(13):2581-90. doi: 10.1084/jem.20111354. Epub 2011 Nov 21. PMID 22110166
- [Background] Jackson PC, Hardwicke J, Bamford A, Nightingale P, Wilson Y, Papini R, Moiemen N. Revised estimates of mortality from the Birmingham Burn Centre, 2001-2010: a continuing analysis over 65 years. Ann Surg. 2014 May;259(5):979-84. doi: 10.1097/SLA.0b013e31829160ca. PMID 23598383
- [Background] Mann EA, Baun MM, Meininger JC, Wade CE. Comparison of mortality associated with sepsis in the burn, trauma, and general intensive care unit patient: a systematic review of the literature. Shock. 2012 Jan;37(1):4-16. doi: 10.1097/SHK.0b013e318237d6bf. PMID 21941222
- [Background] Levy MM, Fink MP, Marshall JC, Abraham E, Angus D, Cook D, Cohen J, Opal SM, Vincent JL, Ramsay G; SCCM/ESICM/ACCP/ATS/SIS. 2001 SCCM/ESICM/ACCP/ATS/SIS International Sepsis Definitions Conference. Crit Care Med. 2003 Apr;31(4):1250-6. doi: 10.1097/01.CCM.0000050454.01978.3B. PMID 12682500
- [Background] Brinkmann V, Reichard U, Goosmann C, Fauler B, Uhlemann Y, Weiss DS, Weinrauch Y, Zychlinsky A. Neutrophil extracellular traps kill bacteria. Science. 2004 Mar 5;303(5663):1532-5. doi: 10.1126/science.1092385. PMID 15001782
- [Background] Mocsai A. Diverse novel functions of neutrophils in immunity, inflammation, and beyond. J Exp Med. 2013 Jul 1;210(7):1283-99. doi: 10.1084/jem.20122220. PMID 23825232
- [Background] Butler KL, Ambravaneswaran V, Agrawal N, Bilodeau M, Toner M, Tompkins RG, Fagan S, Irimia D. Burn injury reduces neutrophil directional migration speed in microfluidic devices. PLoS One. 2010 Jul 30;5(7):e11921. doi: 10.1371/journal.pone.0011921. PMID 20689600
- [Background] Arturson G. Neutrophil granulocyte functions in severely burned patients. Burns Incl Therm Inj. 1985 Jun;11(5):309-19. doi: 10.1016/0305-4179(85)90093-2. PMID 4027746
- [Background] Bjerknes R, Vindenes H, Laerum OD. Altered neutrophil functions in patients with large burns. Blood Cells. 1990;16(1):127-41; discussion 142-3. PMID 2190644
- [Background] Jones CN, Moore M, Dimisko L, Alexander A, Ibrahim A, Hassell BA, Warren HS, Tompkins RG, Fagan SP, Irimia D. Spontaneous neutrophil migration patterns during sepsis after major burns. PLoS One. 2014 Dec 9;9(12):e114509. doi: 10.1371/journal.pone.0114509. eCollection 2014. PMID 25489947
- [Background] The World Health Organisation. Burns [updated April 2014; cited 2015 06.10.2015]. Available from: http://www.who.int/mediacentre/factsheets/fs365/en/.
- [Background] Campisi J. Aging, cellular senescence, and cancer. Annu Rev Physiol. 2013;75:685-705. doi: 10.1146/annurev-physiol-030212-183653. Epub 2012 Nov 8. PMID 23140366
- [Derived] Tullie S, Asiri A, Acharjee A, Moiemen NS, Lord JM, Harrison P, Hazeldine J. Day One Cell-Free DNA Levels as an Objective Prognostic Marker of Mortality in Major Burns Patients. Cells. 2025 Jun 1;14(11):821. doi: 10.3390/cells14110821. PMID 40497997
- [Derived] Hazeldine J, McGee KC, Al-Tarrah K, Hassouna T, Patel K, Imran R, Bishop JRB, Bamford A, Barnes D, Wilson Y, Harrison P, Lord JM, Moiemen NS. Multicentre, longitudinal, observational cohort study to examine the relationship between neutrophil function and sepsis in adults and children with severe thermal injuries: a protocol for the Scientific Investigation of the Biological Pathways Following Thermal Injury-2 (SIFTI-2) study. BMJ Open. 2021 Oct 22;11(10):e052035. doi: 10.1136/bmjopen-2021-052035. PMID 34686556